CLINICAL TRIAL: NCT03198351
Title: Teriflunomide Pregnancy Outcome Exposure Registry: An OTIS Autoimmune Diseases in Pregnancy Project
Brief Title: An Observational Study on Teriflunomide-exposed Pregnancies
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS13499; U1111-1183-8711 (Other: UTN)
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort I: Pregnant women with a confirmed diagnosis of multiple sclerosis (MS) and teriflunomide exposure during the current pregnancy
  Interventions: Drug: Teriflunomide (HMR1726)
- Cohort II: Pregnant women with MS not exposed to teriflunomide during the current pregnancy
- Cohort III: Healthy pregnant women who do not have a known diagnosis of MS and have no known exposure to a known human teratogen
- "Registry" group (not eligible for cohorts): Women who contact the OTIS registry study staff and who do not meet the criteria for the prospective study, for example, at time of contacting the study, having known prenatal diagnosis of congenital defect, or gestation weeks greater than 20 following a first trimester teriflunomide exposure, etc.; these participants will not be included in the primary analysis for the cohort study.

INTERVENTIONS:
Drug: Teriflunomide (HMR1726) — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: Aubagio
  Groups: Cohort I

SUMMARY:
Primary Objective:

To evaluate any potential increase in the risk of major birth defects, in the first year of life, in teriflunomide-exposed pregnancies.

Secondary Objective:

To evaluate the potential effect of teriflunomide-exposure on other adverse pregnancy outcomes including any potential pattern of minor birth defects, spontaneous abortion, stillbirth, preterm delivery, small for gestational age at birth and at 1 year follow-up.

DETAILED DESCRIPTION:
The total study duration per participant is approximately up to 2 years.

* This is a prospective, observational study (no intervention), ie, patient registry.
* The statistical analysis for the cohort study describe baseline characteristics in all three cohorts, and then will compare pregnancy outcomes in cohort 1 to cohort 2 and secondarily to cohort 3.
* For the "registry" group, without comparisons, only descriptive statistics of pregnancy outcomes will be summarized.

ELIGIBILITY:
Inclusion criteria :

* Pregnant women who have provided an oral and/or written consent to enroll no later than 20 completed weeks from last menstrual period (LMP).
* Pregnant women who agree to the conditions and requirements of the study including the interview schedule, release of medical records, and the physical examination of live born infants (up to 1 year post birth).
* Pregnant women with a diagnosis of MS and teriflunomide exposure during pregnancy (Cohort 1).
* Pregnant women with MS but not exposed teriflunomide during pregnancy (Cohort 2).
* Healthy pregnant women who do not have a known diagnosis of MS and have no known exposure to a known human teratogen during pregnancy (Cohort 3).

Exclusion criteria:

* Pregnant women who come in first contact with the project after prenatal diagnosis of a major structural defect (Cohort 1, 2, 3). This does not apply to the "registry" group.
* Pregnant women who first come in contact with the project after 20 completed weeks' gestation (Cohort 1, 2, 3). This does not apply to the "registry" group.
* Pregnant women who had previously enrolled in the study for a previous pregnancy (only 1 pregnancy, per woman, maybe registered) (Cohort 1, 2, 3). This does not apply to the "registry" group.
* Retrospectively reported cases (Cohort 1, 2, 3). This does not apply to the "registry" group.
* Pregnant women with exposures to teriflunomide commencing after the 12th week post-LMP (Cohort 1). This does not apply to the "registry" group.
* Pregnant women who had previously been treated with teriflunomide if they had received any dose of the drug within 2 years prior to the index pregnancy and do not have documented blood levels below 0.02 mcg/mL prior to pregnancy (Cohort 2).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: -Pregnant women will be enrolled at various stages of gestation depending when they are included in the registry; then the pregnant outcome will be followed and for live infants, the follow up will be up to the children's 1 year birthday.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Rate of major structural defects in live born infants | Up to the infant's first year birthday

SECONDARY OUTCOMES:
Proportion of major structural defects in all pregnancies | up to 1 year of age in infant
Specific pattern of 3 or more minor structural defects in live born infants receiving the exam | up to one year after birth
Rate of spontaneous abortion | date of conception to 20 weeks gestation
Rate of preterm delivery | live birth prior to 37 weeks gestation
Proportion of infants who are small for gestational age (less than or equal to the 10th percentile for gestational age and sex) on weight, length, or head circumference | at birth
Proportion of infants less than or equal to the 10th percentile for sex and age on weight, length, or head circumference at 1 year postnatal evaluation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- University of California at San Diego-Site Number:001, San Diego, California, United States
- Investigational Site Number :002, Canada, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org